CLINICAL TRIAL: NCT05000593
Title: Clinical Study of Cord Blood Mononuclear Cells (UCB-MNCs) in the Treatment of Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lili Cao (Other)
Responsible Party: Sponsor-Investigator, Lili Cao, dean of orthopeadic department, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YXLL-KY-2020(040)
Record Dates: First submitted 2020-09-10; First posted 2021-08-11 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Knee Osteoarthritis
Keywords: Cord Blood Mononuclear Cells; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Saline Solution

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- stem cell treating group (Experimental): Intra-articular injection of CB-MNCs (cell count 1×108 cells/time) was performed once every 1 week for a total of 3 times.
  Interventions: Other: normal saline; Other: Cord Blood Mononuclear Cells (UCB-MNCs)

INTERVENTIONS:
Other: normal saline — Intra-articular injection of normal saline
Other: Cord Blood Mononuclear Cells (UCB-MNCs) — Intra-articular injection of Cord Blood Mononuclear Cells (UCB-MNCs)

SUMMARY:
Umbilical cord blood mononuclear cells contain hematopoietic stem cells (HSC), mesenchymal stem cells (MSC), endothelial progenitor cells and other pluripotent stem cells, as well as immature immune cells, which can differentiate into chondrocytes, hematopoietic, epithelial, endothelial and nerve cells. It gives the ability to promote wound healing and vascular microcirculation reconstruction, and has the potential to treat many diseasesHowever, clinical studies on cord blood mononuclear cells in knee osteoarthritis have not been reported in the literature. Therefore, this study aims to explore the safety and effectiveness of cord blood mononuclear cells in the treatment of patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥30 years old, ≤75 years old, no gender limit;
* Meet the KOA diagnostic criteria in the "Classification Criteria for Knee Osteoarthritis" revised by the American College of Rheumatology (ACR);
* According to the X-ray K-L grading and evaluation standard, it is at level II-III;
* Continuous pain for at least 6 months;
* No local or systemic infection;
* There is no obvious contraindication for articular cavity puncture in hematology and biochemical testing;
* Subjects and their families understand the clinical trial protocol and agree to participate in the trial, voluntarily and sign an informed consent form;

Exclusion Criteria:

* Age<30 years old;
* Tumor diseases;
* Severe kidney, lung or liver damage;
* Blood diseases include anemia and thrombocytopenia;
* Type I diabetes;
* Severe effusion;
* Contracture or instability of the knee joint, with an axial deformity greater than 10°;
* Infectious arthritis or skin disease;
* Inject corticosteroids and immunosuppressants into the knee joint within 2 months;
* Suffer from mental illness and poor compliance;
* Cases that the investigator thinks are not suitable for inclusion in the group.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Lysholm score | Compare the changes of 1 month, 3 months, 6 months and one year before treatment (baseline) and after (third injection)
  Evaluation of functional perception of daily activities and motor function levels of different intensities.The score ranges from 0 to 100 points, the lower the score, the more severe the knee joint damage.
American knee society knee score | Compare the changes of 1 month, 3 months, 6 months and one year before treatment (baseline) and after (third injection)
  Evaluation of the overall function and shape of the knee joint.The score ranges from 0 to 100 points. The lower the score, the worse the knee joint function.
the knee injury and osteoarthritis score | Compare the changes of 1 month, 3 months, 6 months and one year before treatment (baseline) and after (third injection)
  A questionnaire for evaluating the effectiveness of knee joint injury and osteoarthropathy treatment based on patient self-assessment management.The KOOS score consists of five parts, and each part contains a different number of questions. Each question has a minimum of 0 points and a maximum of 4 points. After the score of each part is calculated separately, it is converted into a percentile score through the conversion formula. A score of 0 in the converted percentile score means that the function of that part of the joint is extremely poor, and a score of 100 means that the function of this part of the joint is completely normal.
Visual Analog Score for pain | Compare the changes of 1 month, 3 months, 6 months and one year before treatment (baseline) and after (third injection)
  Physicians Global Assessment to measure quality of life.The score ranges from 0 to 10 points, the lower the score, the more severe the pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prieto-Alhambra D, Judge A, Javaid MK, Cooper C, Diez-Perez A, Arden NK. Incidence and risk factors for clinically diagnosed knee, hip and hand osteoarthritis: influences of age, gender and osteoarthritis affecting other joints. Ann Rheum Dis. 2014 Sep;73(9):1659-64. doi: 10.1136/annrheumdis-2013-203355. Epub 2013 Jun 6. PMID 23744977
- [Background] Tang X, Wang S, Zhan S, Niu J, Tao K, Zhang Y, Lin J. The Prevalence of Symptomatic Knee Osteoarthritis in China: Results From the China Health and Retirement Longitudinal Study. Arthritis Rheumatol. 2016 Mar;68(3):648-53. doi: 10.1002/art.39465. PMID 26474054
- [Background] Wang B, Liu W, Xing D, Li R, Lv C, Li Y, Yan X, Ke Y, Xu Y, Du Y, Lin J. Injectable nanohydroxyapatite-chitosan-gelatin micro-scaffolds induce regeneration of knee subchondral bone lesions. Sci Rep. 2017 Dec 1;7(1):16709. doi: 10.1038/s41598-017-17025-6. PMID 29196647
- [Background] McAlindon TE, Bannuru RR, Sullivan MC, Arden NK, Berenbaum F, Bierma-Zeinstra SM, Hawker GA, Henrotin Y, Hunter DJ, Kawaguchi H, Kwoh K, Lohmander S, Rannou F, Roos EM, Underwood M. OARSI guidelines for the non-surgical management of knee osteoarthritis. Osteoarthritis Cartilage. 2014 Mar;22(3):363-88. doi: 10.1016/j.joca.2014.01.003. Epub 2014 Jan 24. PMID 24462672
- [Background] Burke J, Hunter M, Kolhe R, Isales C, Hamrick M, Fulzele S. Therapeutic potential of mesenchymal stem cell based therapy for osteoarthritis. Clin Transl Med. 2016 Dec;5(1):27. doi: 10.1186/s40169-016-0112-7. Epub 2016 Aug 10. PMID 27510262